CLINICAL TRIAL: NCT04161287
Title: Comparison of Efficacy in Stereotactic Body Radiation Therapy (SBRT) of Hepatocellular Carcinoma ≤5 cm With or Without Transcatheter Arterial Chemoembolization (TACE)
Brief Title: Comparison of Efficacy in SBRT of HCC ≤5 cm With or Without TACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JingSun
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-03

CONDITIONS: Small Hepatocellular Carcinoma; Stereotactic Body Radiation Therapy; Transcatheter Arterial Chemoembolization
Keywords: CyberKnife; SBRT; TACE; prognosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SBRT with TACE
  Interventions: Procedure: transcatheter arterial chemoembolization
- SBRT alone

INTERVENTIONS:
Procedure: transcatheter arterial chemoembolization — The hepatocellular carcinoma patients (≤5cm）who received SBRT are devided into two groups: with TACE and SBRT alone.
  Groups: SBRT with TACE

SUMMARY:
The study aims to compare efficacy and adverse reactions of hepatocellular carcinoma participants (≤5cm) who receive stereotactic body radiation therapy with or without transcatheter arterial chemoembolization.The investigators will optimize the combined treatment schedule of SBRT for hepatocellular carcinoma participants by comparing overall survival rates, progression-free survival rates and local control and adverse reaction occurrence rates in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* primary HCC diagnosed by a surgeon and/or radiologist and oncologist according to the international guidelines for the management of HCC or by pathology
* single lesion and longest tumor diameter ≤ 5.0 cm
* CP-A or B classification
* Eastern Cooperative Oncology Group (ECOG) score 0-1;
* distances between tumor and normal organs (esophagus, stomach, duodenum, bowel) are more than 5 mm
* unsuitable for other therapies, such as patients with heart disease, uncontrolled diabetes, uncontrolled hypertension, etc.
* rejecting other therapies such as resection, liver transplantation, etc.
* platelet count≥50 × 109/L, white blood count≥1.5 × 109/L
* patients infected with hepatitis B virus who are treated with adefovir or entecavir; patients infected with hepatitis C virus whose HCV DNA are negative.

Exclusion Criteria:

* tumor thrombus
* lymph node involvement
* extrahepatic metastasis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hepatocellular carcinoma patients whose lesion diameter ≤ 5.0 cm
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2025-01-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival rates | From date of randomization until the date of death from any cause, assessed up to 36 months
  OS is calculated starting from the date of SBRT to the date of the final follow-up or demise of the patients.
Progression-free survival rates | From date of randomization until the date of disease progression or date of death from any cause, whichever came first, assessed up to 36 months
  PFS is estimated starting from the date of SBRT to the date of disease progression or patient death.
Local control rates | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  LC is defined starting from the date of SBRT to the date of treated-lesion progression or patient death.

SECONDARY OUTCOMES:
Radiation-induced liver injury rates | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.
Adverse reaction | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xuezhang Duan, PH.D, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital (Beijing 302 hospital), Beijing, China

REFERENCES:
- [Result] Sun J, Zhang T, Wang J, Li W, Zhang A, He W, Zhang D, Li D, Ding J, Duan X. Biologically effective dose (BED) of stereotactic body radiation therapy (SBRT) was an important factor of therapeutic efficacy in patients with hepatocellular carcinoma (</=5 cm). BMC Cancer. 2019 Aug 28;19(1):846. doi: 10.1186/s12885-019-6063-9. PMID 31455251
- [Result] Zhang T, Sun J, He W, Li H, Piao J, Xu H, Duan X. Stereotactic body radiation therapy as an effective and safe treatment for small hepatocellular carcinoma. BMC Cancer. 2018 Apr 20;18(1):451. doi: 10.1186/s12885-018-4359-9. PMID 29678159
- [Result] Su TS, Lu HZ, Cheng T, Zhou Y, Huang Y, Gao YC, Tang MY, Jiang HY, Lian ZP, Hou EC, Liang P. Long-term survival analysis in combined transarterial embolization and stereotactic body radiation therapy versus stereotactic body radiation monotherapy for unresectable hepatocellular carcinoma >5 cm. BMC Cancer. 2016 Nov 3;16(1):834. doi: 10.1186/s12885-016-2894-9. PMID 27809890
- [Result] Wong TC, Chiang CL, Lee AS, Lee VH, Yeung CS, Ho CH, Cheung TT, Ng KK, Chok SH, Chan AC, Dai WC, Wong FC, Luk MY, Leung TW, Lo CM. Better survival after stereotactic body radiation therapy following transarterial chemoembolization in nonresectable hepatocellular carcinoma: A propensity score matched analysis. Surg Oncol. 2019 Mar;28:228-235. doi: 10.1016/j.suronc.2019.01.006. Epub 2019 Jan 29. PMID 30851906
- [Result] Takayasu K, Arii S, Kudo M, Ichida T, Matsui O, Izumi N, Matsuyama Y, Sakamoto M, Nakashima O, Ku Y, Kokudo N, Makuuchi M. Superselective transarterial chemoembolization for hepatocellular carcinoma. Validation of treatment algorithm proposed by Japanese guidelines. J Hepatol. 2012 Apr;56(4):886-92. doi: 10.1016/j.jhep.2011.10.021. Epub 2011 Dec 13. PMID 22173160